CLINICAL TRIAL: NCT00280995
Title: A Phase 2, Open-Label, Dose Escalation Study to Assess the Safety and Efficacy of ISIS 301012 as Add-on Therapy in Homozygous Familial Hypercholesterolemia Subjects
Brief Title: Dose-escalating Safety Study of ISIS 301012 in Homozygous Familial Hypercholesterolemia Subjects on Lipid Lowering Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kastle Therapeutics, LLC (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Medical Monitor, Genzyme Coporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 301012CS8; EudraCT No.: 2005-004796-38
Record Dates: First submitted 2006-01-20; First posted 2006-01-24 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Hypercholesterolemia, Familial
Keywords: LDL-cholesterol; apoB-100; Homozygous Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Homozygous Familial Hypercholesterolemia | interventions — mipomersen

ARMS (4):
- Cohort A (Experimental): Loading doses followed by weekly maintenance doses
  Interventions: Drug: ISIS 301012
- Cohort B (Experimental): Loading doses followed by weekly maintenance doses
  Interventions: Drug: ISIS 301012
- Cohort C (Experimental): Loading doses followed by weekly maintenance doses
  Interventions: Drug: ISIS 301012
- Cohort D (Experimental): Loading doses followed by extended weekly maintenance doses
  Interventions: Drug: ISIS 301012

INTERVENTIONS:
Drug: ISIS 301012 — 100 mg subcutaneous injections on days 1, 4, 8, 11, 15, 22, 29, and 36
  Arms: Cohort B
Drug: ISIS 301012 — 200 mg subcutaneous injections on days 1, 4, 8, 11, 15, 22, 29, and 36
  Arms: Cohort C
Drug: ISIS 301012 — 300 mg subcutaneous injections on days 1, 4, 8, 11, 15, 22, 29, 36, 43, 50, 57, 64,71, 78, and 85
  Arms: Cohort D
Drug: ISIS 301012 — 50 mg subcutaneous injections on days 1, 4, 8, 11, 15, 22, 29, and 36
  Arms: Cohort A

SUMMARY:
The aim of this study is to assess the safety and efficacy of varying doses of ISIS 301012 as add-on therapy in subjects with Homozygous Familial Hypercholesterolemia

ELIGIBILITY:
Inclusion Criteria:

* Weight ≥ 40 kg for Cohorts A, B, & C; Weight ≥ 50 kg for Cohort D
* Diagnosis of Homozygous Familial Hypercholesterolemia.
* Female must be non-pregnant and non-lactating.
* On stable lipid lowering therapy for at least 4 weeks.
* Lipid values that meet the pre-specified criteria.

Exclusion Criteria:

* Subject had heart problems in the prior 6 months.
* Subject has elevated ALT, AST, or CPK.
* History of renal disease, liver disease, or malignancy.
* Use of oral anticoagulants, unless the dose has been stable for 4 weeks
* Have any other conditions, which in the opinion of the Investigator would make the subject unsuitable for enrollment, or could interfere with the subject participating in or completing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-01; Primary Completion 2007-04 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Percent reduction in LDL-cholesterol from baseline | Week 7 (Cohorts A-C), Week 15 (Cohort D)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (6):
- United States (5):
  - Chicago, Illinois
  - New York, New York
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Houston, Texas
- Amsterdam, Netherlands